CLINICAL TRIAL: NCT03952143
Title: A Prospective, Randomized, Double-Blind Comparison of LY900014 to Insulin Lispro, Both in Combination With Insulin Glargine or Insulin Degludec in Adults With Type 2 Diabetes
Brief Title: A Study of LY900014 Compared to Insulin Lispro (Humalog) in Adults With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16830; I8B-FH-ITSE (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro; Insulin Glargine; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY900014 (Experimental): Participants received 100 units per milliliter (U/mL) LY900014 subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
  Interventions: Drug: LY900014; Drug: Insulin Glargine; Drug: Insulin Degludec
- Insulin Lispro (Active Comparator): Participants received 100 U/mL insulin lispro (Humalog) given SC 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
  Interventions: Drug: Insulin Lispro; Drug: Insulin Glargine; Drug: Insulin Degludec

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro
Drug: Insulin Glargine — Administered SC
Drug: Insulin Degludec — Administered SC

SUMMARY:
The purpose of this study is to see if LY900014 compared to insulin lispro (Humalog), both in combination with insulin glargine or insulin degludec, is safe and effective in participants with type 2 diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have T2D based on the disease diagnostic criteria World Health Organization (WHO) classification.
* Participants must have been treated for at least 90 days prior to screening with either basal insulin + at least 1 prandial injection of bolus insulin or premixed analog/human insulin regimens at least twice daily.
* Participants must be treated no more than 3 oral anti-hyperglycemic medications (OAMs).
* Participants must have a HbA1c ≥7.0% and ≤11.0%.
* Participants must have body mass index (BMI) of ≤35.0 kilograms per meter squared (kg/m2).

Exclusion Criteria:

* Participants must not have been diagnosed, at any time, with type 1 diabetes (T1D) or latent autoimmune diabetes in adults.
* Participants must not have had any episode of severe hypoglycemia within the 6 months prior to screening.
* Participants must not have had 1 or more episodes of diabetic ketoacidosis or hyperglycemic hyperosmolar state within the 6 months prior to screening.
* Participants must not have used thiazolidinediones, glucagon-like peptide 1 (GLP-1) receptor agonist, or pramlintide within 90 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (41):
- Argentina (3):
  - Centro Médico Viamonte, Buenos Aires, AR-C
  - Centro de Investigaciones Metabólicas (CINME), CABA, Buenos Aires
  - Cent Priva Especiali Médicas Ambulatorias Inve Clin CEMAIC, Córdoba
- China (34):
  - Beijing Pinggu District Hospital, Beijing, Cn-11
  - Tianjin Medical University General Hospital, Tianjin, Cn-12
  - Cangzhou People's Hospital, Cangzhou, Cn-13
  - The First Hospital of Qinhuangdao, Qinhuangdao Shi, Cn-13
  - Inner Mongolia People's Hospital, Hohhot, Cn-15
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Cn-21
  - Shengjing Hospital of China Medical University, Shenyang, Cn-21
  - Shanghai Putuo District Center Hospital, Shanghai, Cn-31
  - Shanghai 6th people's hospital, Shanghai, Cn-31
  - The Affiliated Jiangyin Hospital of Southeast University Medical College, Jiangyin, Cn-32
  - Zhongda Hospital Southeast University, Nanjing, Cn-32
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing, Cn-32
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Cn-32
  - The Third Hospital of Nanchang, Nanchang, Cn-36
  - The Central Hospital of Wuhan, Wuhan, Cn-42
  - The First People's Hospital of Yueyang, Yueyang, Cn-43
  - Chongqing General Hospital, Chongqing, Cn-50
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Xingtai People's Hospital, Xingtai, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Qiqihar, Qiqihar, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Wuhan Pu'ai Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Chenzhou NO.1 People's Hospital, Chenzhou, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The First Hospital of Nanjing, Nanjing, Jiangsu
  - China-Japan Union Hospital, CJUH., Changchun, Jilin
  - Siping Central People's Hospital, Siping, Jilin
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Jinan Central Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - Beijing Peking Union Medical College Hospital, Beijing
  - Pingxiang People's Hospital, Pingxiang
- Mexico (4):
  - Unidad de patologia Clinica, Guadalajara, Jalisco
  - Centro de Inv. Medica de Occidente, SC, Zapopan, Jalisco
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Mx-nle
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, N.L.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Compared to Insulin Lispro (Humalog) in Adults With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/6hfa0kzMFqmoyoC8Nn6bXD

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included 8-week lead-in period followed by a 26-week treatment period.
Pre-assignment Details: The purpose of the lead-in period (prior to randomization) was to titrate basal insulin, obtain preliminary diagnostic laboratory tests, and determine baseline hypoglycemia rates. Participants were then randomized into the treatment groups in a 2:1 ratio (LY900014:insulin lispro).
Groups:
- Insulin Lispro (Humalog) Lead-in; Insulin Lispro (Humalog): Participants received 100 units per milliliter (U/mL) insulin lispro (Humalog) subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
- LY900014: Participants received 100 U/mL LY900014 by SC 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
Period: Lead-In Period
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | LY900014
Started | 628 | 0 | 0
Participants Who Received at Least One Dose | 628 | 0 | 0
Completed | 595 | 0 | 0
Not Completed | 33 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Physician Decision | 5 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 0 | 0
Period: Treatment Period
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | LY900014
Started | 0 (Participants received Insulin Lispro during Lead-in Period) | 200 (Participants were randomized to either Insulin lispro or LY900014 in Treatment Period.) | 395 (Participants were randomized to either Insulin lispro or LY900014 in Treatment Period.)
Participants Who Received at Least One Dose | 0 | 200 | 395
Completed | 0 | 191 | 359
Not Completed | 0 | 9 | 36
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 26
Not completed — Due to COVID 19 restrictions | 0 | 2 | 5
Not completed — Participant had taken prohibited concomitant medication | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro (Humalog) | LY900014 | Total
Number analyzed (Participants) | 200 | 395 | 595
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.70 (9.48) | 58.30 (9.26) | 58.50 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 182 | 275
  Male | 107 | 213 | 320
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 11 | 16
  Asian | 162 | 319 | 481
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 53 | 82
  More than one race | 4 | 12 | 16
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 18 | 32 | 50
  China | 162 | 319 | 481
  Mexico | 20 | 44 | 64
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 7.78 (0.88) | 7.73 (0.87) | 7.74 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed model repeated measures (MMRM) model with Baseline + Pooled Country + Number of Bolus at Study Entry Stratum + Type of Basal at Lead-in Stratum + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 26
Population: All randomized Participants with baseline and at least one post-baseline HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 198 | 388
Percentage of HbA1c | -0.63 (0.061) | -0.56 (0.046)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Non-Inferiority — Noninferiority margin = 0.4% for HbA1c; p = 0.321, Mixed Models Analysis; LS Mean Difference = 0.07, 95% CI 2-sided [-0.07 to 0.21]

2. Secondary Outcome: 1-hour Postprandial Glucose (PPG) Excursion During Mixed-Meal Tolerance Test (MMTT)
Description: A standardized MMTT was used to characterize postprandial glucose control following administration of the study insulin. Serum glucose measured at 1-hour timepoint after the start of meal minus fasting serum glucose. Least Squares (LS) mean was determined by analysis of covariance (ANCOVA) model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Number of Bolus at Study Entry Stratum + Type of Basal at Lead-in Stratum + Treatment (Type III sum of squares).
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline 1-hour PPG excursion data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 178 | 326
milligrams per deciliter (mg/dL) | 100.8 (4.00) | 86.2 (3.51)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -14.6, 95% CI 2-sided [-21.9 to -7.4]

3. Secondary Outcome: 2-hour PPG Excursion During MMTT
Description: A standardized MMTT was used to characterize postprandial glucose control following administration of the study insulin. Serum glucose measured at 2-hour timepoint after the start of meal minus fasting serum glucose. Least Squares (LS) mean was determined by analysis of covariance (ANCOVA) model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Number of Bolus at Study Entry Stratum + Type of Basal at Lead-in Stratum + Treatment (Type III sum of squares).
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline 2-hour PPG excursion data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 179 | 327
mg/dL | 133.2 (5.13) | 111.4 (4.47)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -21.8, 95% CI 2-sided [-30.9 to -12.6]

4. Secondary Outcome: Rate of Severe Hypoglycemia
Description: Severe hypoglycemia is defined as an event requiring assistance of another person to administer carbohydrate, glucagon, or other resuscitative actions. Rate of severe hypoglycemia events per 100 years during a defined period was calculated by total number of severe hypoglycemia episodes within the period divided by the cumulative days on treatment from all participants within that treatment group *36525.
Time Frame: Baseline through Week 26
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Events per 100 participant years
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 200 | 395
Events per 100 participant years | 2.00 | 0.52
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Superiority; Relative rate = 0.26, 95% CI 2-sided [0.02 to 2.86]

5. Secondary Outcome: Rate of Documented Symptomatic Postmeal Hypoglycemia
Description: Documented symptomatic postmeal hypoglycemia is an event during which typical symptoms of hypoglycemia are accompanied by blood glucose (BG) of ≤70 mg/dL [3.9 millimole per liter (mmol/L)]. The rate of documented symptomatic postmeal hypoglycemia was estimated by negative binomial model: number of episodes = treatment with log (treatment exposure in days/365.25) as an offset variable
Time Frame: Baseline through Week 26
Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Events per participant per year
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 200 | 395
Events per participant per year
  ≤30 minutes post meal | 0.13 (0.033) | 0.11 (0.020)
  ≤1 hour post meal | 0.25 (0.057) | 0.34 (0.053)
  >1 to ≤2 hours post meal | 0.67 (0.109) | 1.07 (0.145)
  ≤2 hours post meal | 0.92 (0.137) | 1.41 (0.169)
  >2 to ≤4 hours post meal | 1.96 (0.276) | 1.92 (0.214)
  ≤4 hours post meal | 2.89 (0.351) | 3.32 (0.336)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; For ≤30 minutes post meal; Test type: Superiority; Relative rate = 0.90, 95% CI 2-sided [0.49 to 1.66]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014; For ≤ 1 hour post meal; Test type: Superiority; Relative rate = 1.35, 95% CI 2-sided [0.79 to 2.31]
Statistical Analysis 3: Comparison: Insulin Lispro (Humalog) vs LY900014; For >1 to ≤2 hours post meal; Test type: Superiority; Relative rate = 1.60, 95% CI 2-sided [1.06 to 2.42]
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; For ≤2 hours post meal; Test type: Superiority; Relative rate = 1.53, 95% CI 2-sided [1.05 to 2.23]
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014; For >2 to ≤4 hours post meal; Test type: Superiority; Relative rate = 0.97, 95% CI 2-sided [0.69 to 1.39]
Statistical Analysis 6: Comparison: Insulin Lispro (Humalog) vs LY900014; For ≤4 hours post meal; Test type: Superiority; Relative rate = 1.15, 95% CI 2-sided [0.84 to 1.57]

6. Secondary Outcome: Change From Baseline in 1,5-Anhydroglucitol (1,5-AG)
Description: 1,5-anhydroglucitol (1,5-AG) is a marker of short-term glycemic control especially postprandial hyperglycemia. 1,5-AG accurately predicts rapid changes in glycemia and is tightly associated with glucose fluctuations and postprandial glucose. LS Mean was calculated using mixed model repeated measures (MMRM) with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Number of Bolus at Study Entry Stratum + Type of Basal at Lead-in Stratum + Treatment + Time + Treatment*Time (Type III sum of squares)
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline 1,5-AG data.
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 190 | 358
milligram per liter (mg/L) | 2.49 (0.363) | 2.21 (0.280)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; Test type: Superiority; LS Mean Difference = -0.29, 95% CI 2-sided [-1.10 to 0.53]

7. Secondary Outcome: Change From Baseline in 10-Point Self-Monitoring Blood Glucose (SMBG) Values
Description: SMBG 10-point profiles were measured at fasting, 1-hour post morning meal, 2-hours post morning meal, pre midday meal, 1-hour post midday meal, 2-hours post midday meal, pre evening meal, 1-hour post evening meal, 2-hours post evening meal, and bedtime. LS Mean was analyzed using mixed model repeated measures (MMRM) model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Number of Bolus at Study Entry Stratum + Type of Basal at Lead-in Stratum + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline SMBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 170 | 331
mg/dL
  Morning Premeal | 2.2 (2.62) | 4.4 (2.18)
  Morning 1-hour Postmeal: number analyzed (Participants) | 170 | 330
  Morning 1-hour Postmeal | -12.9 (3.77) | -18.1 (3.13)
  Morning 2-hour Postmeal: number analyzed (Participants) | 169 | 329
  Morning 2-hour Postmeal | -15.9 (3.65) | -21.3 (3.02)
  Midday Premeal: number analyzed (Participants) | 167 | 330
  Midday Premeal | -9.8 (3.09) | -5.7 (2.56)
  Midday 1-hour Postmeal: number analyzed (Participants) | 168 | 329
  Midday 1-hour Postmeal | -15.2 (3.52) | -13.9 (2.92)
  Midday 2-hour Postmeal: number analyzed (Participants) | 170 | 328
  Midday 2-hour Postmeal | -24.4 (3.63) | -22.5 (3.02)
  Evening Premeal: number analyzed (Participants) | 169 | 331
  Evening Premeal | -25.0 (3.34) | -10.9 (2.76)
  Evening 1-hour Postmeal: number analyzed (Participants) | 169 | 326
  Evening 1-hour Postmeal | -17.6 (3.65) | -15.6 (3.06)
  Evening 2-hour Postmeal: number analyzed (Participants) | 168 | 325
  Evening 2-hour Postmeal | -22.1 (3.67) | -22.3 (3.05)
  Bedtime: number analyzed (Participants) | 167 | 328
  Bedtime | -22.3 (3.38) | -20.7 (2.82)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; For Morning Premeal; Test type: Superiority; LS Mean Difference = 2.2, 95% CI 2-sided [-2.8 to 7.2]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014; For Morning 1-hour Postmeal; Test type: Superiority; LS Mean Difference = -5.3, 95% CI 2-sided [-12.6 to 2.0]
Statistical Analysis 3: Comparison: Insulin Lispro (Humalog) vs LY900014; For Morning 2-hour Postmeal; Test type: Superiority; LS Mean Difference = -5.4, 95% CI 2-sided [-12.5 to 1.7]
Statistical Analysis 4: Comparison: Insulin Lispro (Humalog) vs LY900014; For Midday Premeal; Test type: Superiority; LS Mean Difference = 4.2, 95% CI 2-sided [-1.8 to 10.1]
Statistical Analysis 5: Comparison: Insulin Lispro (Humalog) vs LY900014; For Midday 1-hour Postmeal; Test type: Superiority; LS Mean Difference = 1.2, 95% CI 2-sided [-5.7 to 8.1]
Statistical Analysis 6: Comparison: Insulin Lispro (Humalog) vs LY900014; For Midday 2-hour Postmeal; Test type: Superiority; LS Mean Difference = 1.9, 95% CI 2-sided [-5.1 to 8.9]
Statistical Analysis 7: Comparison: Insulin Lispro (Humalog) vs LY900014; For Evening Premeal; Test type: Superiority; LS Mean Difference = 14.1, 95% CI 2-sided [7.6 to 20.6]
Statistical Analysis 8: Comparison: Insulin Lispro (Humalog) vs LY900014; For Evening 1-hour Postmeal; Test type: Superiority; LS Mean Difference = 2.0, 95% CI 2-sided [-5.1 to 9.1]
Statistical Analysis 9: Comparison: Insulin Lispro (Humalog) vs LY900014; For Evening 2-hour Postmeal; Test type: Superiority; LS Mean Difference = -0.2, 95% CI 2-sided [-7.3 to 6.8]
Statistical Analysis 10: Comparison: Insulin Lispro (Humalog) vs LY900014; For Bedtime; Test type: Superiority; LS Mean Difference = 1.7, 95% CI 2-sided [-4.7 to 8.1]

8. Secondary Outcome: Change From Baseline in Insulin Dose
Description: LS mean was determined by MMRM model with Baseline + Pooled Country + Hemoglobin A1c Stratum at Baseline + Number of Bolus at Study Entry Stratum + Type of Basal at Lead-in Stratum + Treatment + Time + Treatment*Time (Type III sum of squares)
Time Frame: Baseline, Week 26
Population: All randomized participants with baseline and at least one post-baseline basal insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: Units (U)
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 193 | 369
Units (U)
  Total Daily Insulin Dose | 15.1 (1.13) | 17.8 (0.82)
  Daily Basal Insulin Dose | 0.7 (0.34) | 1.4 (0.26)
  Daily Prandial Insulin Dose | 14.7 (1.04) | 16.7 (0.75)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; For Total Daily Insulin Dose; Test type: Superiority; LS Mean Difference = 2.8, 95% CI 2-sided [0.1 to 5.4]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014; For Daily Basal Insulin Dose; Test type: Superiority; LS Mean Difference = 0.8, 95% CI 2-sided [0.0 to 1.5]
Statistical Analysis 3: Comparison: Insulin Lispro (Humalog) vs LY900014; For Daily Prandial Insulin Dose; Test type: Superiority; LS Mean Difference = 2.0, 95% CI 2-sided [-0.5 to 4.5]

9. Secondary Outcome: Percentage of Participants With HbA1c <7% and ≤6.5%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Only subjects with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Time Frame: Week 26
Population: All randomized participants with baseline and at least one post-baseline HbA1c <7% and ≤6.5% data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Lispro (Humalog) | LY900014
Number analyzed (Participants) | 191 | 358
Percentage of participants
  HbA1c < 7% | 44.50 | 46.65
  HbA1c ≤ 6.5% | 27.23 | 27.93
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog) vs LY900014; For HbA1c < 7%; Test type: Superiority; p = 0.924, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.69 to 1.52]
Statistical Analysis 2: Comparison: Insulin Lispro (Humalog) vs LY900014; For HbA1c ≤6.5%; Test type: Superiority; p = 0.908, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.64 to 1.49]

ADVERSE EVENTS:
Time Frame: Up to 30 weeks
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Insulin Lispro (Humalog): Participants received 100 U/mL insulin lispro (Humalog) subcutaneously (SC) 0-2 minutes before each meal with either basal insulin glargine or insulin degludec given SC once daily.
Arm/Group | Insulin Lispro (Humalog) Lead-in | Insulin Lispro (Humalog) | LY900014
All-Cause Mortality (participants affected / at risk) | 0/628 | 1/200 | 0/395
Serious Adverse Events (participants affected / at risk) | 17/628 | 15/200 | 33/395
Other Adverse Events (participants affected / at risk) | 29/628 | 14/200 | 21/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro (Humalog) Lead-in (N=628) | Insulin Lispro (Humalog) (N=200) | LY900014 (N=395)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 3 (3) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract diabetic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vitreous opacities (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 2 (2) | 0 (0) | 1 (3)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Lispro (Humalog) Lead-in (N=628) | Insulin Lispro (Humalog) (N=200) | LY900014 (N=395)
Upper respiratory tract infection (Infections and infestations) | 29 (31) | 14 (14) | 21 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03952143/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT03952143/SAP_001.pdf